CLINICAL TRIAL: NCT04327492
Title: Clinical, Hematological, and Imagiologic Predictors of Postoperative Complications and Long Term Cardiovascular Events After Carotid Endarterectomy With Regional Anesthesia
Brief Title: Hemathologic and Imagiologic Predictors of Stroke During Carotid Endarterectomy With Regional Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, João Rocha Neves, MD, MSC; MPH, FEBVS, Universidade do Porto
Other Study IDs: 250-19
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Carotid Stenosis; Carotid Endarterectomy
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — blood sample. atherosclerotic plaque
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carotid endarterectomy: This study is a non-interventional prospective cohort study. The population corresponds to patients submitted to CEA under regional anesthesia. Consecutive patients from a tertiary referral center who undergo CEA for carotid artery stenosis (CS) will be prospectively recruited. The expected patient follow-up will be of 5 years.
  The demographics will be recorded in a prospective, protected database. Blood samples will be collected in clot activator serum tubes at three timepoints: timepoint 1 - before surgery (until 15 days before surgery); timepoint 2 up to 48h postoperatively; timepoint
  Interventions: Diagnostic Test: Biomarker - FGF 23; troponin I; PCR - high sensitivity; BNP

INTERVENTIONS:
Diagnostic Test: Biomarker - FGF 23; troponin I; PCR - high sensitivity; BNP — peak wave velocity; gray weale plaque classification

SUMMARY:
Establish and validate biomarkers which improve the predictive value of current risk stratification models for patients benefiting from carotid revascularization, outperform existing biomarkers, and reach clinical application standards.

DETAILED DESCRIPTION:
The authors hypothesize FGF-23 and GDF-15 could predict cerebral ischemia, postoperative complications and long term major cardiovascular events, particularly in patients developing symptomatic neurologic ischemia after circulation shutdown.

Establish and validate biomarkers which improve the predictive value of current risk stratification models for patients benefiting from carotid revascularization, outperform existing biomarkers, and reach clinical application standards.

Clarify the pathophysiology of carotid endarterectomy-related stroke and the role of GDF-15, FGF-23, BNP and hs-troponin I and other biomarkers in the prognosis of symptomatic carotid stenosis.

Imagiologic markers are to be included - intima-media; gray weale plaque classification, cerebral CT Peak wave velocity

ELIGIBILITY:
Inclusion Criteria:

- consecutive patients from a tertiary referral center who undergo CEA for carotid artery stenosis (CS) under regional anesthesia

Exclusion Criteria:

* general anesthesia
* carotid stenting

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients selected and submited to carotid endarterectomy under regional anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 272 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Stroke | 30 days, long-term
Clavien dindo>3 | 30 days, long-term
MACE | 30 days, long-term
  AMI, stroke, Major adverse limb event, acute hear faillure hospitalization, all cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Joao R Neves, MD, MSC, MPH, Principal Investigator — Universidade do Porto
Locations (1):
- Faculdade de Medicina da Universidade do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No